CLINICAL TRIAL: NCT05777681
Title: Management of Aorto-iliac Infection With BioIntegral Surgical No-React® Bovine Pericardial Xenografts
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Tshomba Yamume, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5142
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Aortic Diseases
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Aortic Surgery — open surgical repair with resection of infected aortic segment, debridement of surrounding tissue and in situ graft replacement.

SUMMARY:
Aortic infections (AIs), including aortic graft infections (AGI) as well as mycotic aortic aneurysms (MAA), are rare. The aim of this study is to present our experience with xenogeneic aortic and aortoiliac reconstructions using the BioIntegral Surgical No-React® bovine pericardial graft.

ELIGIBILITY:
Inclusion Criteria:

* Aortic infection
* Mycotic Aneurysm
* Aortic Graft Infection

Exclusion Criteria:

* Absence of signs of infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent replacement of an infected aneurysm or graft with a BioIntegral Surgical No-React® bovine pericardial prosthesis at our Institution.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Early Mortality | 30 days
  Mortality 30 days after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No